CLINICAL TRIAL: NCT01754649
Title: Assessment of Use of Misoprostol to Facilitate the Insertion of Intrauterine Contraceptives After Failure of Insertion. A Randomized Double-blind Clinical Trial
Brief Title: Use of Misoprostol in Case of Insertion Failure of Intrauterine Contraceptives
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Luis Bahamondes (Other)
Responsible Party: Sponsor-Investigator, Luis Bahamondes, PI, University of Campinas, Brazil
Organization: University of Campinas, Brazil (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Unicamp/2012/LB
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Cervical Stenosis
Keywords: intrauterine device; insertion failure
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- misoprostol vaginal 200 mcg (Active Comparator): The study group will receive two doses of misoprostol (200mcg each tablet) vaginal 12 and 4 hours prior insertion After 24 hours of the insertion failure the women will return to the clinic and a new attempt of insertion will be done. At this time we will evaluate if the insertion was able to do or not.
  Interventions: Drug: Misoprostol
- placebo (Placebo Comparator): The placebo group will receive two doses of placebo vaginal 12 and 4 hours prior insertion. After 24 hours of the insertion failure the women will return to the clinic and a new attempt of insertion will be done. At this time we will evaluate if the insertion was able to do or not.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — The study group will receive two doses of misoprostol (200mcg each tablet) vaginal 12 and 4 hours prior insertion. After 24 hours of the insertion failure the women will return to the clinic and a new attempt of insertion will be done. At this time we will evaluate if the insertion was able to do or not.
  Other Names: PROSTOKOS

SUMMARY:
To assess the usefulnes sof misoprostol versus placebo (in a double-blind placebo controlled randomized clinical trial)to facilitate the insertion of copper-IUD and the levonorgestrel-releasing intrauterine system (LNG-IUS) in cases of failure due to cervical stenosis in either nulligravidas and parous women. Additionally to evaluate the side-effects of the misoprostol. The hypothesis is that misoprostol may be better than placebo.

DETAILED DESCRIPTION:
Women attended at the Family Planning clinic of the University of Campinas who requested the insertion of a copper-IUD or an LNG-IUS and who failed in the attempt due to cervical stenosis will be randomized in two groups (1:1). The study group will receive two doses of misoprostol (200mcg each tablet) vaginal 12 and 4 hours prior insertion and the control group will receive placebo in the same schedule. The sample will be 50 women in each group. After 24 hours of the insertion failure the women will return to the clinic and a new attempt of insertion will be done. At this time we will evaluate if the insertion was able to do or not. The data will be analyzing with χ2 test for independent samples. After that a multiple logistic analysis will be perform to evaluate the associated variables with the result (failure or successful) insertion. The level of significance will be established at P<.005.

ELIGIBILITY:
Inclusion Criteria:

Women aged > 18 and <50 years old; Requesting insertion of and IUD or an LNG-IUS Failure of IUD insertion

Exclusion Criteria:

Refuse to participate Lost to follow-up at the return visit

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
ease of insertion of intrauterine contraceptives | 12 months
  The study group will receive two doses of misoprostol (200mcg each tablet) vaginal 12 and 4 hours prior insertion and the control group will receive placebo in the same schedule. The sample will be 50 women in each group. After 24 hours of the insertion failure the women will return to the clinic and a new attempt of insertion will be done. At this time we will evaluate if the insertion was able to do or not.

SECONDARY OUTCOMES:
Side-effects of misoprostol | 12 months
  To assess the side-effects of misoprostol versus placebo

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Family Planning Clinic, University of Campinas, Campinas, São Paulo
  - University of Campinas, Campinas, São Paulo

REFERENCES:
- [Derived] Bahamondes MV, Espejo-Arce X, Bahamondes L. Effect of vaginal administration of misoprostol before intrauterine contraceptive insertion following previous insertion failure: a double blind RCT. Hum Reprod. 2015 Aug;30(8):1861-6. doi: 10.1093/humrep/dev137. Epub 2015 Jun 3. PMID 26040478